CLINICAL TRIAL: NCT00619138
Title: A Randomized, Controlled Study of a Stepped-care Model for the Treatment of Social Phobia and Panic Disorder in Adults
Brief Title: Treatment of Social Phobia and Panic Disorder in Adults
Acronym: TSPPA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Odd E Havik, professor, Haukeland University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17650
Record Dates: First submitted 2008-01-16; First posted 2008-02-20 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Social Phobia; Panic Disorder
Keywords: Cognitive therapy; Stepped care; Self-help; Internet; Anxiety
MeSH Terms: conditions — Phobia, Social; Panic Disorder; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Behavioral: individual cognitive-behavioural therapy
- 2 (Active Comparator)
  Interventions: Behavioral: stepped care model

INTERVENTIONS:
Behavioral: individual cognitive-behavioural therapy — 1 session per week for 12 weeks
  Arms: 1
Behavioral: stepped care model — three steps: short psycho-education, a 10 weeks Internet-based self-help program, 12 weeks individual cognitive-behavioural therapy
  Arms: 2

SUMMARY:
The purpose of this study is to compare a stepped care model for the treatment of social phobia and panic disorder with standard psychological treatment. The stepped care model comprises three steps: short psycho-education, a 10 weeks Internet-based self-help program, 12 weeks individual cognitive-behavioural therapy. Patients are assessed at each step and taken out of the study if they show significant clinical improvement and follow for 12 months. Patients are randomized to either the stepped care model or standard psychological treatment, i.e. individual cognitive-behavioural therapy. All treatment components are manualized.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnoses of panic disorder or social phobia
* Informed consent

Exclusion Criteria:

* Alcohol/drug dependency
* Major depressive disorder
* Psychosis
* Unstable medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2008-03; Primary Completion 2012-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Clinical Severity Ratings | End of treatment and 12 months follow-up

SECONDARY OUTCOMES:
Questionnaires: The Panic Attack Scale The Body Sensations Questionnaire The Agoraphobic Cognitions Questionnaire The Mobility Inventory for Agoraphobia Social Phobia Scale The Social Interaction Anxiety Scale | End of treatment and 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: odd e havik, PhD, Principal Investigator — University of Bergen
Locations (1):
- haukelandUH, Bergen, Norway

REFERENCES:
- [Derived] Haug T, Nordgreen T, Ost LG, Tangen T, Kvale G, Hovland OJ, Heiervang ER, Havik OE. Working alliance and competence as predictors of outcome in cognitive behavioral therapy for social anxiety and panic disorder in adults. Behav Res Ther. 2016 Feb;77:40-51. doi: 10.1016/j.brat.2015.12.004. Epub 2015 Dec 11. PMID 26708332
- [Derived] Haug T, Nordgreen T, Ost LG, Kvale G, Tangen T, Andersson G, Carlbring P, Heiervang ER, Havik OE. Stepped care versus face-to-face cognitive behavior therapy for panic disorder and social anxiety disorder: Predictors and moderators of outcome. Behav Res Ther. 2015 Aug;71:76-89. doi: 10.1016/j.brat.2015.06.002. Epub 2015 Jun 9. PMID 26081010